CLINICAL TRIAL: NCT01941927
Title: Phase II Clinical Trial of the MEK Inhibitor Trametinib With the AKT Inhibitor GSK2141795 in BRAF Wild-type Melanoma
Brief Title: Trametinib With GSK2141795 in BRAF Wild-type Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adil Daud (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor-Investigator, Adil Daud, Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13855; NCI-2013-01849 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2013-08-30; First posted 2013-09-13 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Melanoma
Keywords: Melanoma; Wild-type; BRAF
MeSH Terms: conditions — Melanoma | interventions — trametinib; GSK2141795

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trametinib, GSK2141795 (Experimental): Trametinib (GSK1120212)
  * Oral
  * 2 mg
  * Daily
  * Number of Cycles: until progression or unacceptable toxicity develops
  GSK2141795
  * Oral
  * 25 mg
  * Daily
  * Number of Cycles: until progression or unacceptable toxicity develops
  Interventions: Drug: Trametinib (GSK1120212); Drug: GSK2141795

INTERVENTIONS:
Drug: Trametinib (GSK1120212) — Trametinib is a highly selective allosteric inhibitor of MEK1 and MEK2 activation and kinase activity.
  Other Names: MEKINIST
Drug: GSK2141795 — GSK 2141795 is an ATP competitive subnanomolar pan-AKT inhibitor. In order to measure the true potency of GSK 2141795, potency (Ki*) values were determined in a filter binding assay using lower enzyme concentrations (0.1, 0.7, and 0.2 nM for human AKT1, AKT2, and AKT3, respectively). Using a sandwich ELISA, GSK 2141795 inhibited phosphorylation of GSK-3β in BT474 and LNCaP cell lines with EC50 values of 143 and 34 nM, respectively. Since phosphorylation of GSK-3β can be modulated by other enzymes (PKA, PKC, and RSK),cellular activity of GSK 2141795 was evaluated using a phospho-PRAS40 ELISA. GSK 2141795 inhibited the phosphorylation of PRAS40 with EC50 values of 39 and 55 nM for BT474 and LNCaP cells, respectively.

SUMMARY:
This is a multicenter phase II clinical study of trametinib in combination with GSK2141795 in patients with BRAF wild-type mutation melanoma. All patients will receive continuous dosing of trametinib (2 mg) in combination with GSK2141795 (25 mg) oral daily until progression of disease, withdrawal of consent, or the development of intolerable treatment associated toxicity. Imaging (CT or MRI) will be performed within 7 days prior to day 1 of Odd Cycles, starting with Cycle 3.

Patients may continue treatment with trametinib in combination with GSK2141795 on trial until disease progression or the development of unacceptable toxicity that does not improve with maximal supportive care or dose reduction per protocol.

Treatment-associated adverse events will be assessed based on clinical and laboratory findings using the Common Toxicity Criteria for Adverse Events, version 4.0. Adverse event (AE) assessments will be performed every week through cycle 3 day 1, and on day 1 for every cycle thereafter. AEs and Serious adverse events (SAE)s will be monitored by UCSF's Data Safety Monitoring Committee.

Safety assessments will include medical history, physical examination, Complete Blood Count (CBC) with differential, chemistries panel, thyroid function and pregnancy tests, ECGs, and ophthalmology evaluations. Screening assessments will also include a transthoracic echocardiogram or multiple-gated acquisition (MUGA) scan, and brain imaging.

It is estimated that 48 patients will complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically or cytologically confirmed Malignant Melanoma.
3. Unresectable Stage III or Stage IV disease.
4. Measureable disease by RECIST 1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
6. Resolution of all acute toxic effects of prior radiotherapy, chemotherapy or surgical procedures to NCI CTCAE Version 4.0 grade ≤1. At least 2 weeks must have elapsed since the end of prior systemic treatment, radiotherapy, or major surgical procedure.
7. Evidence of tumor DNA showing either NRAS mutation or NRAS Wild-Type (WT)/BRAF WT. BRAF genotype must be determined by a CLIA-approved assay. NRAS genotyping may be determined by Sanger sequencing, melting point polymerase chain reaction (PCR) assay, Sequenome, or NextGen sequencing.
8. Adequate Bone Marrow and Organ function as defined:

   * Hemoglobin ≥ 9 g/dL
   * Absolute neutrophil count ≥ 1,500/mm3
   * Platelet count ≥ 100,000/mm3
   * Bilirubin ≤ 1.5 times normal limit
   * aspartate aminotransferase (AST) /alanine aminotransferase (ALT) ≤ 5 times the upper limit of normal if liver metastasis present or ≤2.5 X upper limit of normal (ULN) if no liver metastases are present.
   * Creatinine ≤ 2 mg/dL

Exclusion Criteria:

1. Progressive central nervous system (CNS) metastatic disease. Patients with CNS metastases are allowed only if previously treated and stable for 8 weeks or more, and patient is neurologically intact off steroids. The stability must be documented by MRI/CT over a period of 8 weeks or greater.
2. Congestive Heart Failure with significant limitation of activity New York Heart Association (NYHA) class III or IV
3. Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
4. QTc >480 mSec , unless presence of bundle branch block. In this case, observed QTc - (QRS-150) should be ≤ 480 msec.
5. More than 1 prior chemotherapy regimen. Patients may have had any prior immunotherapy regimens but must be at least 6 weeks out from anti-CTLA4 or anti-PD-1 antibody treatment and show progression based on immune response evaluation criteria.
6. Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy and for 4 months following last dose.
7. Prior treatment with any AKT or MEK inhibitor
8. Retinal or Fundal disease (including macular degeneration, retinal vein occlusion, hypertensive or diabetic retinopathy).
9. Inflammatory Bowel Disease, malabsorption syndrome or diarrhea > Grade 1.
10. Need for treatment with drugs that are known potent CYP3A inhibitors. Current use or anticipated need for treatment with drugs that are known potent CYP3A or CYP1A2 inducers.
11. Prior malignancy will be allowed as long as the patient is known to be free of disease for at least 5 years. Prior Squamous cell carcinoma (SCC), Basal Cell, cervical cancer, early stage prostate cancer, ductal carcinoma in situ (DCIS) or melanoma (second primary) are allowed even if <5 years from diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09-10 (Actual); Primary Completion 2014-10-14 (Actual); Study Completion 2017-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil Daud, M.D., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Algazi AP, Esteve-Puig R, Nosrati A, Hinds B, Hobbs-Muthukumar A, Nandoskar P, Ortiz-Urda S, Chapman PB, Daud A. Dual MEK/AKT inhibition with trametinib and GSK2141795 does not yield clinical benefit in metastatic NRAS-mutant and wild-type melanoma. Pigment Cell Melanoma Res. 2018 Jan;31(1):110-114. doi: 10.1111/pcmr.12644. Epub 2017 Nov 2. PMID 28921907

RESULTS

PARTICIPANT FLOW:
Groups:
- NRAS Wildtype: Patients without NRAS (neuroblastoma RAS viral oncogene homolog) exon 1 and 2 mutations
- NRAS Mutant: Patients with NRAS exon 1 and 2 mutations (NRAS mutant) identified by Sanger sequencing or exon-capture next-generation sequencing
Period: Overall Study
Arm/Group | NRAS Wildtype | NRAS Mutant
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with NRAS exon 1 and 2 mutations (NRAS mutant) identified by Sanger sequencing or exon-capture next-generation equencing and patients without these mutations (wild-type (WT)). The sample size for each arm was based on a Simon 2-stage stage design.
Groups:
- NRAS Wildtype: Patients without NRAS exon 1 and 2 mutations
- Total: Total of all reporting groups
Arm/Group | NRAS Wildtype | NRAS Mutant | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Mean (Full Range); unit: years] | 59.3 [40 to 86] | 56.8 [19 to 67] | 58.5 [19 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 8 | 7 | 15
Eastern Cooperative Oncology Group (ECOG) status: 0 [Count of Participants; unit: Participants] — Participants were rated using the ECOG Performance Status Scale. Status had to be 0 to 2 in order to be eligible for the study.
  Grade 0: Normal activity. Fully active, able to carry on all pre-disease performance without restriction
  Grade 1: Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work)
  Grade 2: In bed < 50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours
  Participants
    ECOG status 0 | 6 | 2 | 8
    ECOG status 1 | 4 | 8 | 12
    ECOG status 2 | 0 | 0 | 0
Stage [Count of Participants; unit: Participants] — Histological confirmation of Malignant Melanoma using the American Joint Committee on Cancer (AJCC) tumor/node/metastasis (TNM) classification and staging system.
  M1a: Metastases to skin, soft tissue (including muscle), and/or nonregional lymph nodes
  M1b: Lung metastasis, with or without M1a involvement
  M1c: Distant metastasis to non-central nervous system (CNS) visceral sites with or without M1a or M1b involvement
  Participants
    M1a | 0 | 2 | 2
    M1b | 0 | 2 | 2
    M1c | 10 | 6 | 16
Lactate Dehydrogenase (LDH) level [Count of Participants; unit: Participants]
  LDH normal | 2 | 2 | 4
  LDH elevated | 8 | 8 | 16
Genotype [Count of Participants; unit: Participants]
  Genotype NRAS Q61H | 0 | 1 | 1
  Genotype NRAS Q61K | 0 | 3 | 3
  Genotype NRAS Q61L | 0 | 1 | 1
  Genotype NRAS Q61R | 0 | 5 | 5
  BRAF Wild Type (WT) /NRAS WT | 10 | 0 | 10
Subtype [Count of Participants; unit: Participants]
  Cutaneous | 6 | 0 | 6
  Mucosal | 0 | 8 | 8
  Acral | 1 | 2 | 3
  Uveal | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Only those participants who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response These participants will have their response classified according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) method, where the baseline target lesion sum of longest diameter (LD) will be used as reference by which to characterize the objective tumor response. An objective response is defined as an overall response of complete response (CR), partial response (PR), or stable disease (SD) with a confirmatory scan or evaluation at time of final disease response determination.
Time Frame: Up to 2 years from beginning of therapy
Population: Reported here are a number of participants that achieved the best objective response defined as stable disease
Measure: Count of Participants; unit: Participants
Arm/Group | NRAS Wildtype | NRAS Mutant
Number analyzed (Participants) | 10 | 10
Participants | 5 | 4

2. Secondary Outcome: Progression-Free Survival of Patients Treated With the Combination of Trametinib and GSK 2141795
Description: Time from randomization to objective tumor progression or death. Participants who die without documentation of disease progression and before it was time to conduct the first tumor reassessment, will be considered inevaluable or not assessed adequately
Time Frame: Up to 2 years from beginning of therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NRAS Wildtype | NRAS Mutant
Number analyzed (Participants) | 10 | 10
months | 2.8 [2.6 to 2.9] | 2.3 [2.1 to 2.5]

3. Secondary Outcome: Overall Survival of Patients Treated With the Combination of Trametinib and GSK 2141795
Time Frame: Up to 2 years from beginning of therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NRAS Wildtype | NRAS Mutant
Number analyzed (Participants) | 10 | 10
months | 3.5 [0.6 to 6.4] | 4 [0.9 to 7]

4. Secondary Outcome: Time-to-Progression (TTP) of Patients Treated With the Combination of Trametinib and GSK 2141795
Description: Time from treatment initiation until objective tumor progression observed. Only those participants who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response. Participants who exhibit objective disease progression prior to the end of Cycle 1 will be considered evaluable. Response will also be considered inevaluable for any participants receiving treatment (regardless of how much was received) who did not have any follow-up assessment completed before initiation of alternative treatment or participants who die without documentation of disease progression and before it was time to conduct the first tumor reassessment, will be considered inevaluable or not assessed adequately
Time Frame: Up to 2 years from beginning of therapy
Population: The drug combination failed to produce objective responses in participants with either NRAS mutant or NRAS wild-type melanoma in TTP evaluable patient population. No objective responses for progression in TTP specific evaluable participants population were observed so endpoint could not be calculated.
Arm/Group | NRAS Wildtype | NRAS Mutant
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Severe Adverse Events (Grade 3 and 4) Reported by Patients Related With the Treatment of Trametinib and GSK2141795.
Time Frame: Up to 2 years from beginning of therapy
Measure: Number; unit: Severe Adverse Events
Arm/Group | Trametinib, GSK2141795
Number analyzed (Participants) | 10
Severe Adverse Events | 6

ADVERSE EVENTS:
Time Frame: Patient toxicity will be collected from time of first treatment at weekly scheduled study visits. Patients will be followed for toxicity for 30 days after last dose of study drug or removal from study, or until death, whichever occurs first. Patients removed from study for unacceptable treatment related adverse event(s) will be followed additionally until resolution or stabilization of all treatment related adverse events to Grade 2 or lower
Groups:
- Trametinib, GSK2141795: Trametinib (GSK1120212)
  * Oral, 2 mg Daily
  * Number of Cycles: until progression or unacceptable toxicity develops
  GSK2141795
  * Oral, 25 mg Daily
  * Number of Cycles: until progression or unacceptable toxicity develops
Arm/Group | Trametinib, GSK2141795
All-Cause Mortality (participants affected / at risk) | 12/20
Serious Adverse Events (participants affected / at risk) | 5/20
Other Adverse Events (participants affected / at risk) | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trametinib, GSK2141795 (N=20)
diarrhea (Gastrointestinal disorders) | 1
failure to thrive (General disorders) | 1
decubitus ulcer (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trametinib, GSK2141795 (N=20)
Diarrhea (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 2
Anal fistula (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 4
Fever (General disorders) | 3
Chills (General disorders) | 1
Malaise (General disorders) | 1
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Sinus pain (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Rash pustular (Infections and infestations) | 2
Bladder infection (Infections and infestations) | 1
Alkaline phosphatase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No